CLINICAL TRIAL: NCT06391281
Title: The Effect of Fistula Education Given to Patients Receiving Hemodialysis Treatment on Self-Care Behaviors
Brief Title: Effect of Fistula Training in Hemodialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kırklareli University (Other)
Responsible Party: Principal Investigator, Özlem Özdemir, Dr. lecturer, Kırklareli University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Kirklareli Ozlem Ozdemir
Record Dates: First submitted 2024-04-24; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Hemodialysis
Keywords: hemodialysis; Fistula; self care; education
MeSH Terms: conditions — Fistula | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): routine care
- Education (Experimental): The patient receiving hemodialysis treatment will be given fistula self-care training in 2 sessions. An educational booklet will be provided after the training.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The patient receiving hemodialysis treatment will be given fistula self-care training in 2 sessions. An educational booklet will be provided after the training.And routine care
  Other Names: experimental
  Arms: Education

SUMMARY:
It was planned to examine the effect of fistula-related education given to patients receiving hemodialysis treatment on their self-care behaviors.

Nurse-led education about fistula for hemodialysis patients affects fistula self-care behaviors.

Nurse-led training regarding fistula to hemodialysis patients does not affect fistula self-care behaviors.

DETAILED DESCRIPTION:
Hemodialysis patients in the experimental group will be given face-to-face training in 2 sessions. Patients will also receive an educational brochure on fistula self-care. Simultaneously, patients will receive routine treatment and care.

No intervention will be performed on patients in the control group. These patients will receive normal treatment and care.

A pre-test will be applied to both groups at the first meeting and their self-care behaviors related to fistula will be examined. Three months later, fistula-related self-care behaviors will be evaluated again with the relevant scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,with chronic kidney disease
* Having a fistula as a vascular access route
* Receiving hemodialysis treatment for at least 6 months

Exclusion Criteria:

* Those with acute renal failure,
* Having a graft and catheter as a vascular access route,
* Not volunteering to participate in the research
* Those with communication problems (hearing, language, understanding, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-04-26 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Patient Information Form | 1-3 month
  Contains disease-related and sociodemographic information
Self-Care Behavior Assessment Scale Regarding Arteriovenous Fistula in Hemodialysis Patients | 1-3 month
  he scale was adapted from Sousa et al. Developed by. Turkish validity and reliability, İkiz et al. It was done by. The scale consists of the subscales "management of symptoms and signs" and "prevention of complications". An increase in the score indicates that the person's self-care behaviors regarding fistula care are improving